CLINICAL TRIAL: NCT03623503
Title: Clinical Criteria for a Pathogen in Term Newborn Suspected of Neonatal Sepsis
Acronym: IMF-NN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-18- PrTourneux
Record Dates: First submitted 2018-08-02; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Newborn Sepsis
Keywords: newborn; neonatal spesis; clinical sriteria
MeSH Terms: conditions — Neonatal Sepsis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- first group: Observational study of 25 newborn with a likely EOS
  Interventions: Other: Observational study
- second group: Observational study of v33 newborn with a possible EOS
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study

SUMMARY:
Neonatal early onset sepsis (EOS) diagnosis is difficult due to lack of sensivity and specificity markers. The investigators conduced a restrospectif study to all term born infants born between 1 january and 31 December 2013 and hospitalized for suspect EOS. The presence of neonatal symptoms at birth appears to be a useful clinical marker of probable neonatal EOS.

DETAILED DESCRIPTION:
neonatal early onset spesis (EOS) remains animportant etiology of neonatal morbidity and mortality. Neonatal early onset sepsis (EOS) diagnosis is difficult due to lack of sensivity and specificity markers. Diagnosis is difficults due to lack of sensivity and specificity markers. The investigators conduced a restrospectif study to all term born infants born between 1 january and 31 December 2013 and hospitalized for suspect EOS.The objective of the study was to identify early clinical signs in newborn infants with suspected neonatal sepsis to differentiate a likely infection with pathogen bacteria in the gastric suction culture.The presence of neonatal symptoms at birth appears to be a useful clinical marker of probable neonatal EOS.

ELIGIBILITY:
Inclusion Criteria:

* Children born at the University Hospital Center in Amiens between 1 January and 31 December 2013 and hospitalized in the neonatology department for suspicion of MFIs

Exclusion Criteria:

* Child born before 37 weeks of amenorrhea and / or having a failure in the birth room requiring immediate transfer to neonatal resuscitation or intensive care neonatology

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children born between 1 January and 31 December 2013 and hospitalized in the neonatology department for suspicion of MFIs.
  Presence of early clinical signs, ie before 72 hours of life.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-02-21 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
clinical signs in newborn infants | 1 year
  The objective of the study was to determine early clinical signs in newborn infants with suspected neonatal sepsis to differentiate a likely infection with pathogen bacteria in gastric suction culture.The investigators conduced a retrospective study and all term newborn infant born between 1 january and 31 december 2013 and hospitalized for suspected EOS were included.From the computerized medical file, which is filled in exhaustively, the data were given in the form of continuous values or in the form of a category: maternal age, gestationality, delivery period, delivery method, childbirth administration of maternal antibiotherapy. the parameters at birth were recorded in the same way: sex of the newborn, measurements of birth (birth weight, height, cranial perimeter).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Tourneux, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No